CLINICAL TRIAL: NCT03316872
Title: Pembrolizumab and Stereotactic Radiotherapy Combined in Subjects With Advanced Hepatocellular Carcinoma - A Phase II Study
Brief Title: Study of Pembrolizumab and Radiotherapy in Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to the shift in systemic treatment paradigm for HCC precluding further enrolment.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEMRAD
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab and Stereotactic Body Radiotherapy (SBRT) (Experimental): Pembrolizumab, intravenously, at a dose of 200 mg, once every 3 weeks
  SBRT starting Day 2 of Cycle 1 of pembrolizumab treatment, given in 5 fractions over 10-15 days.
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: KEYTRUDA
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT involves delivery of high doses of radiation therapy in smaller fractions

SUMMARY:
This is a phase 2 study whose purpose is to assess the efficacy of the combination of pembrolizumab and stereotactic body radiotherapy (SBRT) in patients with advanced hepatocellular carcinoma (HCC) who have experienced disease progression after treatment with sorafenib.

DETAILED DESCRIPTION:
Pembrolizumab will be administered intravenously as a 30-minute infusion at a dose of 200 mg every 21 days, until disease progression or intolerable toxicity.

Stereotactic radiotherapy will commence on day 2 of the first cycle of pembrolizumab, and will be delivered in 5 fractions over 8-15 days in accordance with institutional protocol.

Subjects will be re-evaluated for response every 12 weeks. In addition to a baseline scan, confirmatory scans should also be obtained 4-8 weeks following initial documentation of objective response.

Response and progression will be evaluated in this study using both RECIST 1.1and (iRECIST) guideline (Seymor 2017).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial
* Be ≥18 years of age on day of signing informed consent.
* Have a histologically- or cytologically-confirmed diagnosis of hepatocellular carcinoma (HCC), and at least one measurable lesion.
* Have current liver function meeting Child Pugh Class A (5-6 points), with no encephalopathy or ascites.
* Have intrahepatic HCC amenable to stereotactic body radiotherapy (SBRT):
* maximum 10 lesions to be treated, and
* total tumor diameter to be treated <20 cm
* No single liver tumor >15 cm in diameter
* No evidence of common or main branch bile duct invasion
* No evidence of direct tumor extension into stomach, duodenum, small bowel, large bowel or diaphragm
* Smaller satellites of HCC or non-definite HCC need not be encompassed within SBRT volumes if needed to respect normal tissue limits.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have demonstrated disease progression, after previous treatment with sorafenib for advanced or metastatic disease, lasting a minimum of 8 week period, allowing for appropriate interruptions and dose reductions.
* Have recovered (to ≤ grade 1) from prior toxicities related to previous treatments at the time of study enrollment, with the exception of alopecia or skin depigmentation.
* Be tested during screening for Hepatitis B-Virus surface antigen (HbsAg) status. Patients may be included in the study if they have adequately controlled hepatitis B
* Patients must be tested during study screening for hepatitis C virus (HCV) RNA status. Patients with chronic infection by HCV who are untreated are allowed on study. In addition, patients with successful HCV treatment are allowed as long as 4 weeks have passed between completion of HCV therapy and start of study treatment.
* Demonstrate adequate organ function.
* Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential. Men treated or enrolled on this trial must agree to use adequate contraception prior to and for 4 months after completion of pembrolizumab administration.

Exclusion Criteria:

* Has received any second-line systemic therapy for advanced HCC after disease progression following sorafenib therapy, or has had prior radiotherapy to the proposed treatment field.
* Is currently participating and receiving experimental treatment as part of a clinical trial, or has participated in a study of an immune checkpoint inhibitor and received study therapy, or used an investigational device within 4 weeks of the first dose of treatment.
* Has had a previous solid organ transplant, a diagnosis of immunodeficiency, or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has liver tumor not amenable to SBRT, or has had prior upper abdominal radiation therapy within planned volumes (exceeding standard tolerances).
* Has a histological or cytological diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma-HCC.
* Has had prior radioembolization or other selective internal radiotherapy treatment to the liver.
* Has dual active HBV infection (HBsAg (+) and/or detectable HBV DNA) and HCV infection (anti-HCV Ab(+) and detectable HCV RNA) at study entry.
* Has had esophageal or gastric variceal bleeding within 3 months prior to study enrollment.
* Has had encephalopathy in the past 6 months, or has clinically apparent ascites at the time of study enrollment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known history of prior invasive malignancy except if the subject has undergone curative-intent therapy with no evidence of disease recurrence for 2 years prior to study entry. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, low-risk prostate cancer or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* HHas active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy at a dose of ≤ 10 mg/day of prednisone or equivalent) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has alcohol related or non-alcoholic steatohepatitis (NASH) related cirrhosis.
* Has had a history of significant active or unstable heart disease
* Has received a live vaccine or live-attenuated vaccine within 30 days of planned start of study therapy. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J. Knox, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 patients of a planned 22 were enrolled
Groups:
- Pembrolizumab and Stereotactic Body Radiotherapy (SBRT): Pembrolizumab, intravenously, at a dose of 200 mg, once every 3 weeks
  SBRT starting Day 2 of Cycle 1 of pembrolizumab treatment, given in 5 fractions over 10-15 days.
  Pembrolizumab: Pembrolizumab is a humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Stereotactic Body Radiotherapy (SBRT): SBRT involves delivery of high doses of radiation therapy in smaller fractions
Period: Overall Study
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
Started | 18
Completed | 17 (Of the 18 patients included, 17 were evaluable for response)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Of the 18 patients included, 17 were evaluable for response.
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 66.5 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5
  White | 12
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  Canada | 18
Number of participants with history of liver disease [Count of Participants; unit: Participants]
  Hep B | 3
  Hep C | 6
  MASLD/Alcohol/other | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To assess the systemic efficacy of combined SBRT and pembrolizumab in subjects with advanced HCC who have experienced disease progression after previous therapy, as measured by overall response rate (ORR).
Time Frame: 3 years
Population: Patients with histologically confirmed advanced HCC with a Childs-Pugh score of 5 or 6 and ECOG 0-1 were eligible. Patients must have progressed on one line of prior TKI therapy for advanced HCC. Patients had to have intrahepatic HCC, treatable with personalized SBRT (27.5 Gy to 50 Gy in 5 fractions). A maximum of 10 hepatic lesions could be treated with a total sum of tumor diameters <20cm, with no limit on the extent of MVI (as long as it could be encompassed with SBRT.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 17
percentage of participants | 41 [18 to 67]

2. Secondary Outcome: Progression-free Survival
Description: To determine the progression-free survival (PFS), in subjects receiving combination treatment with pembrolizumab and SBRT for advanced HCC who have experienced disease progression after sorafenib therapy.
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (Full Range); unit: years
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 17
years | 0.45 [0.233 to 0.825]

3. Secondary Outcome: Overall Survival Rate
Description: To determine the overall survival (OS) in subjects receiving combination treatment with pembrolizumab and SBRT for advanced HCC who have experienced disease progression after sorafenib therapy.
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (Full Range); unit: years
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 17
years | 1.05 [0.475 to 2.15]

ADVERSE EVENTS:
Time Frame: 3 years, up to 36 months
Description: Adverse Events were recorded from the time of screening until 30 days after last dose.
  Adverse events (AEs) and treatment related adverse events (TRAEs) were recorded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Arm/Group | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 14/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT) (N=18)
Blood bilirubin increased grade 2 (Investigations) | 3 (3)
Blood bilirubin increased grade 1 (Investigations) | 1 (1)
Blood bilirubin increased grade 3 (Investigations) | 1 (1)
Acute kidney injury grade 3 (Renal and urinary disorders) | 1 (1)
Tumor lysis syndrome grade 3 (Metabolism and nutrition disorders) | 1 (1)
Ascites grade 3 (Gastrointestinal disorders) | 4 (5)
Aspartate aminotransferase increased grade 3 (Investigations) | 2 (2)
Febrile neutropenia grade 3 (Blood and lymphatic system disorders) | 1 (1)
RASH grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Generalized muscle weakness grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial fibrillation grade 1 (Cardiac disorders) | 1 (1)
Hepatic failure grade 4 (Hepatobiliary disorders) | 1 (1)
Hepatic failure grade 5 (Hepatobiliary disorders) | 1 (1)
Pneumonitis grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Myocarditis grade 4 (Cardiac disorders) | 1 (1)
Myocarditis grade 5 (Cardiac disorders) | 1 (1)
Alanine aminotransferase increased grade 3 (Investigations) | 2 (2)
MOUTH SORES grade 2 (General disorders) | 1 (1)
Fever grade 1 (General disorders) | 1 (1)
Acidosis grade 4 (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia grade 2 (Metabolism and nutrition disorders) | 1 (1)
Vomiting grade 2 (Gastrointestinal disorders) | 1 (1)
Dyspnea grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills grade 1 (General disorders) | 1 (1)
Anorexia grade 2 (Metabolism and nutrition disorders) | 1 (1)
Flu like symptoms grade 1 (General disorders) | 1 (1)
Cough grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancreatitis grade 3 (Gastrointestinal disorders) | 1 (1)
Bone infection grade 3 (Infections and infestations) | 2 (3)
Seizure grade 4 (Nervous system disorders) | 1 (1)
Cardiac arrest grade 4 (Cardiac disorders) | 1 (1)
Cardiac arrest grade 5 (Cardiac disorders) | 1 (1)
Respiratory failure grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthritis grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
AML grade 2 (Blood and lymphatic system disorders) | 1 (1)
Edema limbs grade 2 (General disorders) | 1 (1)
Anemia grade 4 (Blood and lymphatic system disorders) | 1 (1)
Upper gastrointestinal hemorrhage grade 3 (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Stereotactic Body Radiotherapy (SBRT) (N=18)
Diarrhea grade 1 (Gastrointestinal disorders) | 7 (9)
Diarrhea grade 2 (Gastrointestinal disorders) | 2 (2)
Anorexia grade 1 (Metabolism and nutrition disorders) | 5 (6)
Anorexia grade 2 (Metabolism and nutrition disorders) | 5 (5)
Anorexia grade 3 (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased grade 1 (Investigations) | 12 (30)
Aspartate aminotransferase increased grade 2 (Investigations) | 7 (15)
Aspartate aminotransferase increased grade 3 (Investigations) | 3 (5)
Alkaline phosphatase increased grade 1 (Investigations) | 11 (19)
Alkaline phosphatase increased grade 2 (Investigations) | 3 (7)
Alanine aminotransferase increased grade 1 (Investigations) | 10 (22)
Alanine aminotransferase increased grade 2 (Investigations) | 5 (7)
Alanine aminotransferase increased grade 3 (Investigations) | 3 (3)
Colitis grade 1 (Gastrointestinal disorders) | 1 (1)
Hypotension grade 1 (Vascular disorders) | 1 (1)
Hypotension grade 3 (Vascular disorders) | 1 (1)
Creatinine increased grade 1 (Investigations) | 3 (5)
Fatigue grade 1 (General disorders) | 9 (13)
Fatigue grade 2 (General disorders) | 9 (12)
Insomnia grade 2 (Psychiatric disorders) | 1 (1)
Abdominal distension grade 1 (Gastrointestinal disorders) | 1 (1)
Constipation grade 1 (Gastrointestinal disorders) | 6 (9)
Constipation grade 2 (Gastrointestinal disorders) | 1 (1)
Constipation grade 3 (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased grade 1 (Investigations) | 7 (20)
Blood bilirubin increased grade 2 (Investigations) | 6 (11)
Blood bilirubin increased grade 3 (Investigations) | 3 (5)
Rash maculo-papular grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration grade 2 (Investigations) | 1 (1)
Dehydration grade 3 (Investigations) | 1 (1)
Hyponatremia grade 1 (Metabolism and nutrition disorders) | 5 (16)
Hyponatremia grade 3 (Metabolism and nutrition disorders) | 4 (6)
Ascites grade 1 (Gastrointestinal disorders) | 1 (1)
Ascites grade 2 (Gastrointestinal disorders) | 5 (5)
Ascites grade 3 (Gastrointestinal disorders) | 1 (1)
Abdominal pain grade 1 (Gastrointestinal disorders) | 9 (9)
Abdominal pain grade 2 (Gastrointestinal disorders) | 5 (6)
Abdominal pain grade 3 (Gastrointestinal disorders) | 1 (2)
Edema limbs grade 1 (General disorders) | 4 (4)
Edema limbs grade 2 (Gastrointestinal disorders) | 3 (3)
Hypertension grade 1 (Vascular disorders) | 1 (1)
Hypertension grade 2 (Vascular disorders) | 3 (3)
Chest pain grade 1 (Cardiac disorders) | 1 (1)
Breast pain grade 1 (Reproductive system and breast disorders) | 1 (1)
Platelet count decreased grade 1 (Investigations) | 11 (20)
Platelet count decreased grade 2 (Investigations) | 6 (10)
Platelet count decreased grade 3 (Investigations) | 3 (3)
Chest wall pain grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Purpura grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Gynecomastia grade 1 (Reproductive system and breast disorders) | 1 (1)
INR increased grade 1 (Investigations) | 5 (9)
Hypocalcemia grade 1 (Metabolism and nutrition disorders) | 7 (20)
Hypocalcemia grade 2 (Metabolism and nutrition disorders) | 4 (7)
White blood cell decreased grade 1 (Investigations) | 5 (17)
White blood cell decreased grade 2 (Investigations) | 3 (11)
White blood cell decreased grade 3 (Investigations) | 2 (3)
Hypothyroidism grade 2 (Endocrine disorders) | 1 (1)
Neutrophil count decreased grade 1 (Investigations) | 2 (8)
Neutrophil count decreased grade 2 (Investigations) | 4 (5)
Neutrophil count decreased grade 3 (Investigations) | 2 (3)
Cough grade 1 (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Cough grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Lymphocyte count decreased grade 1 (Investigations) | 6 (13)
Lymphocyte count decreased grade 2 (Investigations) | 9 (20)
Lymphocyte count decreased grade 3 (Investigations) | 9 (14)
Lymphocyte count decreased grade 4 (Investigations) | 1 (2)
Hypoalbuminemia grade 1 (Investigations) | 7 (26)
Hypoalbuminemia grade 2 (Investigations) | 4 (8)
Hypoalbuminemia grade 3 (Investigations) | 1 (1)
Hypomagnesemia grade 1 (Metabolism and nutrition disorders) | 6 (15)
Anemia grade 1 (Blood and lymphatic system disorders) | 9 (17)
Anemia grade 2 (Blood and lymphatic system disorders) | 5 (20)
Anemia grade 3 (Blood and lymphatic system disorders) | 4 (7)
Pain grade 1 (General disorders) | 3 (4)
Pain grade 2 (General disorders) | 1 (2)
Pain grade 3 (General disorders) | 1 (1)
Pain in extremity grade 1 (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity grade 2 (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity grade 3 (Musculoskeletal and connective tissue disorders) | 2 (2)
Vomiting grade 1 (Gastrointestinal disorders) | 3 (4)
Vomiting grade 2 (Gastrointestinal disorders) | 2 (2)
Vomiting grade 3 (Gastrointestinal disorders) | 1 (1)
Dizziness grade 1 (Nervous system disorders) | 2 (2)
Dehydration grade 2 (Metabolism and nutrition disorders) | 1 (1)
Dehydration grade 3 (Metabolism and nutrition disorders) | 1 (1)
Pruritus grade 1 (Skin and subcutaneous tissue disorders) | 6 (9)
Pruritus grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
PRURIGO NODULES grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain grade 2 (Musculoskeletal and connective tissue disorders) | 1 (2)
Lymph node pain grade 1 (Blood and lymphatic system disorders) | 1 (1)
Localized edema grade 1 (General disorders) | 1 (1)
Pancreatitis grade 3 (Gastrointestinal disorders) | 1 (1)
Neck pain grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain grade 1 (General disorders) | 1 (1)
Non-cardiac chest pain grade 2 (General disorders) | 1 (1)
Dyspnea grade 1 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea grade 2 (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increased grade 1 (Investigations) | 1 (1)
Lipase increased grade 4 (Investigations) | 1 (2)
Weight loss grade 1 (Investigations) | 1 (1)
Weight loss grade 2 (Investigations) | 1 (1)
Pleural effusion grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia grade 3 (Metabolism and nutrition disorders) | 1 (1)
Myalgia grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung infection grade 2 (Infections and infestations) | 2 (2)
Arthritis grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
LIVER PAIN grade 1 (Hepatobiliary disorders) | 1 (1)
Glucose intolerance grade 2 (Metabolism and nutrition disorders) | 1 (1)
Pneumonitis grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu like symptoms grade 1 (General disorders) | 2 (2)
Flu like symptoms grade 2 (General disorders) | 1 (1)
Dyspepsia grade 2 (Gastrointestinal disorders) | 2 (2)
Nausea grade 1 (Gastrointestinal disorders) | 6 (8)
Nausea grade 2 (Gastrointestinal disorders) | 5 (6)
Gastrointestinal pain grade 1 (Gastrointestinal disorders) | 1 (1)
Sinus bradycardia grade 1 (Cardiac disorders) | 1 (1)
JOINT STIFFNESS grade 1 (Musculoskeletal and connective tissue disorders) | 1 (2)
Dysgeusia grade 1 (Nervous system disorders) | 1 (1)
Dysgeusia grade 2 (Nervous system disorders) | 1 (2)
REGURGITATION grade 1 (Gastrointestinal disorders) | 1 (1)
Malaise grade 1 (General disorders) | 1 (1)
Dysphagia grade 1 (Gastrointestinal disorders) | 1 (1)
Sneezing grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infarction grade 3 (Cardiac disorders) | 1 (1)
Adrenal insufficiency grade 2 (Endocrine disorders) | 2 (2)
Pain (General) grade 1 (General disorders) | 1 (1)
Hyperglycemia grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia grade 2 (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia grade 3 (Metabolism and nutrition disorders) | 2 (2)
TSH INCREASED grade 1 (Investigations) | 1 (1)
RASH TO ARMS BILATERALLY grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
JOINT PAIN grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash acneiform grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Chills grade 1 (General disorders) | 1 (1)
Edema face grade 1 (General disorders) | 1 (1)
Gastroesophageal reflux disease grade 2 (Gastrointestinal disorders) | 2 (2)
Confusion grade 1 (Psychiatric disorders) | 1 (1)
Anxiety grade 1 (Psychiatric disorders) | 1 (1)
Dry mouth grade 1 (Gastrointestinal disorders) | 1 (1)
HEAT RASH grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
URINARY TRACT PAIN grade 1 (Renal and urinary disorders) | 1 (1)
Oral pain grade 1 (Gastrointestinal disorders) | 1 (1)
LACTATE DEHYDROGENASE INCREASED grade 1 (Investigations) | 1 (1)
Fever grade 1 (General disorders) | 2 (2)
Irritability grade 1 (General disorders) | 1 (1)
Hepatic failure grade 3 (Hepatobiliary disorders) | 1 (1)
Acute kidney injury grade 1 (Renal and urinary disorders) | 2 (2)
Acute kidney injury grade 3 (Renal and urinary disorders) | 1 (1)
Sepsis grade 4 (Infections and infestations) | 1 (1)
Cataract grade 3 (Eye disorders) | 1 (1)
Bloating grade 1 (Gastrointestinal disorders) | 1 (1)
Bloating grade 2 (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged grade 1 (Investigations) | 1 (2)
Hypophosphatemia grade 2 (Metabolism and nutrition disorders) | 4 (7)
Hypophosphatemia grade 3 (Metabolism and nutrition disorders) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hiccups grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucosal infection grade 1 (Infections and infestations) | 1 (1)
Joint effusion grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision grade 1 (Eye disorders) | 1 (1)
Nasal congestion grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event grade 1 (Vascular disorders) | 1 (1)
BLOOD TRANSFUSION grade 2 (General disorders) | 1 (1)
Photosensitivity grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma grade 1 (Vascular disorders) | 1 (1)
Toothache grade 2 (Gastrointestinal disorders) | 1 (1)
Bruising grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Dry skin grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Dry eye grade 1 (Eye disorders) | 1 (1)
RHINORRHEA grade 1 (General disorders) | 1 (1)
Sore throat grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03316872/Prot_SAP_000.pdf